CLINICAL TRIAL: NCT06512870
Title: Can Near Infrared Spectroscopy (NIRS) or Intramuscular Glucose Monitoring (IMGM) Detect Impaired Perfusion in the Anterior Compartment of the Leg in Patients With Tibial Fractures? "Proof of Concept" Pilot Study
Brief Title: Can Near-Infrared Spectroscopy (NIRS) or Intramuscular Glucose Levels Detect Impaired Leg Compartment' Perfusion?
Acronym: NIRS
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202400236
Record Dates: First submitted 2024-04-30; First posted 2024-07-22 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Compartment Syndromes
Keywords: ACS (Acute compartment syndrome); NIRS (near infrared spectroscopy); IM (intramuscular) glucose
MeSH Terms: conditions — Compartment Syndromes | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Known ACS: Patients, aged 18 to 75 years, with diagnosis of unilateral tibial fracture, complicated by Acute Compartment syndrome and/or acute vascular compromise (leg ischemia, absent pulses below the knee), as diagnosed and confirmed by ED physician, orthopedic surgeon and/or vascular surgeon. Only patients with depth to anterior compartment <2.5 cm as measured by the ultrasound will be enrolled.
  Interventions: Diagnostic Test: Near infrared spectroscopy (NIRS)

INTERVENTIONS:
Diagnostic Test: Near infrared spectroscopy (NIRS) — A technique that relies on differential absorption of infrared light to provide relative estimation of tissue oxygenation, has been successfully used to monitor perfusion of various tissues, including muscle tissue of the lower extremity.

SUMMARY:
Near infrared spectroscopy (NIRS), a technique that relies on differential absorption of infrared light to provide relative estimation of tissue oxygenation, has been successfully used to monitor perfusion of various tissues, including muscle tissue of the lower extremity, however available research reports mixed success and this technology is not currently a standard of care for patients with leg fractures.

The investigators propose use of NIRS technology in patients with diagnosis of tibial fracture and acute compartment syndrome to detect / document impaired perfusion of the anterior compartment of the leg, as compared to their non-broken leg. The investigators also propose measurement of intramuscular glucose level in the affected leg and compare it to a fingerstick glucose to detect relative hypoglycemia in the affected muscular compartment. If proven effective, NIRS, or IM glucose, or both techniques could be used for clinical monitoring of patients with tibial fractures at risk for acute compartment syndrome.

DETAILED DESCRIPTION:
Inclusion criteria:

* Patient's age: 18 - 75 years old
* Diagnosis of tibial fracture or fracture-dislocation with diagnosis of acute compartment syndrome AND/OR diagnosis of concomitant vascular injury with documented loss of pulses in the leg below the knee
* Unilateral injury (i.e. only one leg is affected)
* Depth of anterior compartment of the leg < 2.5 cm (as measured by ultrasound) Study size - 7-10 patients

Procedure of enrollment:

When diagnosis of tibial fracture with vascular compromise or established ACS is made by the ED physician and confirmed by the Orthopedic surgeon, study team will be notified immediately (by the orthopedic service).

Study team member will approach the study candidate, explain the purpose of the study and obtain the informed consent.

After obtaining the consent, pre-scanning of the anterior compartment of the leg will be performed at bedside to measure the depth between the surface of the skin and the muscle.

If depth of the anterior muscular compartment found to be <2.5 cm, NIRS sensors will be applied to the skin of the broken leg at that location, and to the corresponding location on the uninjured leg. Sensors will be connected to the monitor and readings will be obtained until patient enters the OR.

Sensor will be removed from the skin of the injured extremity, but will stay in place on uninjured leg to describe tissue perfusion changed which occur during anesthesia.

When incision is made by the surgeon, upon entering the anterior muscular-fascial compartment, blood sample will be obtained from the cut surface of the muscle for glucose concentration measurement. At the same time fingerstick will be performed and capillary glucose will be measured. Both glucose readings will be recorded.

Before entering the anterior compartment, intracompartmental pressure measurement will be performed by the surgeon using a sterile arterial line catheter attached to the transducer connected to the anesthesia monitor, or with the Striker device - at surgeon discretion.

At completion of the surgery, sensor will be re-applied on the anterior compartment of the injured leg before dressing application.

Monitoring of both extremities will continue for 72 hrs following surgery, (if condition of the operative extremity permits presence of the sensor).

All available data stored in the monitor then will be downloaded and analyzed. (Please see more specific time points below).

Data analysis:

NIRS readings will be collected at the following time=points:

* "time 0" (after sensors' application) - both legs
* "Time in the OR - surgery" - for uninjured leg only - 1 hr after induction of general anesthesia
* "Time in the OR - post surgery", after emergence from anesthesia - both legs
* Every 6 hrs thereafter for the first 24 hrs,
* Every 12 hrs for subsequent 48 hrs. Graphic analysis: Superimposed graphs (trajectories) of all patients in each group (with vascular injury and without vascular injury).

Means will be calculated for the injured and uninjured leg for all time points as mentioned above.

Graphs for means will be also created and analyzed. Additionally, the following data will be collected: demographic data ( patient's age, gender), fracture diagnosis, time from admission to surgery, type of surgery performed (external temporary fixation, internal fixation with intramedullary nail vs with plate(s)).

Data will be downloaded to the encrypted thumb-drive and transferred to a password-protected electronic file on HSC server. Only HRRC-approved investigators will have access to the files.

After completion of the study all electronic data will be destroyed. Temporary data sheets will be used to facilitate data collection. They will be stored in the locked cabinet in the Anesthesiology department offices, away from patient areas.

Upon enrollment patients will be given numbers from 1 to 10. After complete set of data is obtained, each patient will be de-identified. Should need arise to refer back to the electronic data, patients will be only identified by their numbers (from 1 to 10) and their respective sets of data.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age to 75 years of age
2. Diagnosis of tibial fracture or fracture-dislocation complicated by diagnosis of acute compartment syndrome AND/OR diagnosis of concomitant vascular injury with documented loss of pulses in the leg below the knee
3. Unilateral injury (i.e. only one leg is affected)

5) Depth of anterior compartment of the leg < 2.5 cm (as measured by ultrasound) 6) Willing to consent to the study

Exclusion Criteria:

1. Younger than 18 years of age or over 75 years of age
2. Skin damage, open wound or infection at the skin overlying the anterior muscular compartment, preventing NIRS sensor placement.
3. Depth to the muscle more than 3 cm as assessed with ultrasound.
4. History of fasciotomy performed on the affected leg.
5. Inability to obtain the informed consent from the patient of legal guardian or healthcare surrogate.
6. Language barrier- Inability to read or understand spoken English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to UF Hospital with diagnosis of unilateral tibial fractures, complicated by acute compartment syndrome and/or acute vascular compromise of the fractures leg.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Use of NIRS to detect changes in perfusion in tibial fractures with acute compartment syndrome or leg ischemia due vascular compromise. | 72 hours
  NIRS sensors will be applied to the skin overlying anterior compartment of the injuries and uninjured legs. Uninjured leg will serve as a control leg. Readings from both legs will be recorded continuously until patient enters OR for emergent surgery. At that point NIRS sensor will be removed to allow skin prep for surgical procedure. NIRS sensor will be re-applied to the skin at the completion of the surgery before leg is wrapped with the dressing. Monitoring of both extremities will be continued for 72 hours.
  If NIRS readings of the affected extremity will be reliably lower as compared to unaffected extremity, and that difference will reverse after surgery (fasciotomy), where NIRS reading of the affected extremity should be at least equal to or, most likely, higher than those of the unaffected extremity, that will prove that NIRS monitoring can be used to detect acute compartment syndrome and muscular ischemia.
Use of point-of-care IM glucose to document relative hypoglycemia in the anterior compartment of the affected leg as an indicator of ACS and/or tissue ischemia. | once, intraoperatively
  When incision is made by the surgeon, upon entering the anterior muscular-fascial compartment, surgeon will obtain small drop of blood (by aspiration with a 2 ml syringe from the cut surface of the muscle) and pass it on to the study personnel to apply it onto the test strip for glucose measurement. At the same time fingerstick will be performed and capillary glucose will be measured. Both glucose readings will be recorded.
  If intramuscular glucose readings in the affected extremity show relative hypoglycemia, i.e. glucose in the affected compartment will be lower than the fingerstick performed at the hand at the same time, that will prove that intramuscular glucose monitoring can be used to detect acute compartment syndrome and muscular ischemia.

CONTACTS AND LOCATIONS:
Locations (1):
- UF Health, Gainesville, Florida, United States